CLINICAL TRIAL: NCT05093634
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial: Multiple Independent Sub-studies of Setmelanotide in Patients With POMC/PCSK1, LEPR, NCOA1(SRC1), or SH2B1 Gene Variants in the Melanocortin-4 Receptor Pathway
Brief Title: EMANATE: A Study of Setmelanotide in Patients With Specific Gene Variants in the MC4R Pathway
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-035
Record Dates: First submitted 2021-09-30; First posted 2021-10-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Genetic Obesity
Keywords: Melanocortin-4 Receptor Pathway; Genetic Obesity; Hunger; Hyperphagia; POMC; PCSK1; LEPR; SH2B1; NCOA1 (SRC1)
MeSH Terms: conditions — Obesity; Hyperphagia | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- POMC or PCSK1 variant (Experimental): 1:1 Randomization
  Interventions: Drug: Setmelanotide; Drug: Placebo
- LEPR variant (Experimental): 1:1 Randomization
  Interventions: Drug: Setmelanotide; Drug: Placebo
- NCOA1 (SRC1) variant (Experimental): 1:1 Randomization
  Interventions: Drug: Setmelanotide; Drug: Placebo
- SH2B1 variant (Experimental): 1:1 Randomization
  Interventions: Drug: Setmelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — Subcutaneous Injection
Drug: Placebo — Subcutaneous Injection

SUMMARY:
The protocol describes a randomized, double-blind, placebo-controlled trial with independent sub-studies of setmelanotide in patients with obesity and at least one of the specific gene variants in the Melanocortin-4 Receptor pathway:

* POMC or PCSK1 (Sub-study 035a)
* LEPR (Sub-study 035b)
* SRC1 (Sub-study 035c)
* SH2B1 (Sub-study 035d)

The objectives and endpoints are identical for these sub-studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pre-identified:

  * Heterozygous genetic variant in the POMC gene or PCSK1 gene
  * Heterozygous genetic variant in the LEPR gene
  * Homozygous, heterozygous, or compound heterozygous variant in the NCOA1 (SRC1)
  * Homozygous, heterozygous, or compound heterozygous variant in SH2B1 gene, or chromosomal 16p11.2 deletion encompassing the SH2B1 gene
* Between 6 and 65 years of age at the time of provision of informed consent/assent
* Obesity, defined as BMI ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th percentile for age and gender for patients 6 up to 17 years of age
* Patient and/or parent or guardian is able to understand and comply with the requirements of the study and is able to understand and sign the written informed consent/assent
* Patient and/or parent or guardian reports that patient experienced childhood obesity, defined as the patient and/or parent or guardian reporting that the patient was significantly overweight during childhood
* Agree to use a highly effective form of contraception throughout the study and for 90 days following the study
* Reported history of lifestyle intervention of diet and exercise
* Reported history of hyperphagia

Key Exclusion Criteria:

* Weight loss of 2% or greater in the previous 3 months
* Recent history of bariatric surgery
* Significant psychiatric disorder(s)
* Suicidal ideation, attempt or behavior
* Clinically significant pulmonary, cardiac, endocrine/metabolic, hepatic or oncologic disease
* Glycated hemoglobin (HbA1C) >10% at Screening
* History of significant liver disease or severe kidney disease
* History or close family history (parents or siblings) of melanoma, or patient history of oculocutaneous albinism
* Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion)
* Participation in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing
* Previously enrolled in a clinical study involving setmelanotide or any previous exposure to setmelanotide
* Significant hypersensitivity to any excipient in the study drug
* If female, pregnant or breastfeeding

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in mean change in body weight in patients treated with setmelanotide compared to placebo, assessed as percent change in BMI | Baseline to 52 weeks

SECONDARY OUTCOMES:
The proportion of patients who achieve at least 5% reduction in BMI in patients treated with setmelanotide compared to placebo | Baseline to 52 weeks
The difference in mean change in body weight in adult patients treated with setmelanotide compared to placebo, assessed as percent change in baseline body weight | Baseline to 52 weeks
The difference in mean percent change in the weekly average most hunger score in patients treated with setmelanotide compared to placebo | Baseline to 52 weeks
The proportion of patients who achieve at least 10% reduction in BMI in patients treated with setmelanotide compared to placebo | Baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (56):
- United States (32):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - HonorHealth Bariatric Center, Scottsdale, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Advent Health, Altamonte Springs, Florida
  - InQuest Medical Research, Suwanee, Georgia
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Metro Detroit Endocrinology Center, Dearborn, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - Metropolitan Hospital Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Ten's Medical Center - Pediatric Endocrinology Clinic, Staten Island, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Montefiore, Pittsburgh, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Texas Tech, Amarillo, Texas
  - Texas Children's Hospital, Houston, Texas
  - Biopharma Informatic, Houston, Texas
  - Rio Grande Valley Endocrine Center, McAllen, Texas
  - Endocrine Associates of Dallas and Plano, Plano, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
  - Marshfield Clinic Research Foundation, a Division of Marshfield Clinic, Inc, Marshfield, Wisconsin
- University of Alberta - Alberta Diabetes Institute (ADI), Edmonton, Alberta, Canada
- France (5):
  - GH Est Hopital Femme Mere Enfant, Lyon
  - Hu Pitie Salpetriere Aphp, Paris
  - Hopital Armand Trousseau, Paris
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Pessac
  - Hôpital Félix Guyon Bellepierre, Saint-Denis
- Germany (4):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Endokrinologikum Frankfurt, Frankfurt
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Ulm, Ulm
- University of Patras School of Medicine, Rio, Greece
- Israel (2):
  - Hasharon Hospital, Petah Tikva
  - Chaim Sheba MC, Safra Children's Hospital, Ramat Gan
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- University of Puerto Rico, San Juan, Puerto Rico
- Spain (4):
  - Hospital Sant Joan de Deu, Barcelona, Barcelona
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria de Málaga, Málaga
  - Hospital General de Valencia, Valencia
- United Kingdom (5):
  - Bristol Royal Hospital for Children, Bristol
  - University of Cambridge, Cambridge
  - Aintree University Hospital, Liverpool
  - London Medical - The London Diabetes Centre, London
  - University College London Hospitals NHS Foundation Trust, London